CLINICAL TRIAL: NCT05080699
Title: Effect of Hypocaloric, High-protein Enteral Formula on Body Weight and Health Outcomes in Obese HEN Patients: A Pilot Study
Brief Title: Evaluating Benefit of Peptide Based Diet in Obese HEN Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-012322
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Tube feeding; Obesity; Body mass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peptamen Intense in obese home enteral nutrition patients after stroke (Experimental): Subjects currently enrolled in Mayo Clinic Home Enteral Nutrition (HEN) program and anticipated to require tube feedings to provide 90% or more of feeding needs will be placed on a Peptamen Intense VHP for up to 12 weeks.
  Interventions: Dietary Supplement: Peptamen Intense VHP, Nestlé Health Science, Switzerland

INTERVENTIONS:
Dietary Supplement: Peptamen Intense VHP, Nestlé Health Science, Switzerland — An enteral formula containing hydrolyzed whey protein, maltodextrin, long-chain triglycerides, medium chain triglycerides (MCT), vitamins and minerals. Compared to standard enteral formula, Peptamen Intense is higher in protein (37 kcal%) and lower in carbohydrates (29 kcal%). The energy content is 1.0 kcal/mL.

SUMMARY:
The purpose of this study is to assess the effects of a low energy, high protein tube feeding formula on body weight in tube fed patients who are obese. It will also assess study formula tolerance as well as impact of the study formula on lean body mass, blood pressure, blood sugar and lipids.

ELIGIBILITY:
Inclusion Criteria:

* Home Enteral Nutrition (HEN) patient receiving at least 90% of energy needs from enteral nutrition.
* BMI > 30.
* History of stroke.
* Weight stable over the past month.

Exclusion Criteria:

* Diagnosis of cancer undergoing active treatment (chemotherapy, radiation, immunotherapy).
* Life expectancy of less than 6 months.
* Stage IV or higher kidney disease (GFR < 30).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline, 3 months
  Change in body weight, measured in kg

SECONDARY OUTCOMES:
Change in lean body mass | Baseline, 12 weeks
  Change in lean body mass, measured as the difference between total body weight and body fat weight reported in percentage
Change in systolic and diastolic blood pressure | Baseline, 12 weeks
  Change in systolic and diastolic blood pressure, measured in mmHg
Change in HbA1c | Baseline, 12 weeks
  Change in hemoglobin A1c, measured in percentage
Change in c-peptide | Baseline, 12 weeks
  Change in c-peptide serum levels, measured in ng/mL
Change in total cholesterol | Baseline, 12 weeks
  Change in total cholesterol, measured in milligrams (mg) of cholesterol per deciliter (dL) of blood.
Change in HDL | Baseline, 12 weeks
  Change in HDL, measured in milligrams (mg) of HDL per deciliter (dL) of blood.
Change in LDL | Baseline, 12 weeks
  Change in LDL, measured in milligrams (mg) of LDL per deciliter (dL) of blood.
Change in triglycerides | Baseline, 12 weeks
  Change in triglycerides, measured in milligrams (mg) of triglycerides per deciliter (dL) of blood.
Change in percent goal calories provided with enteral nutrition | Baseline, 12 weeks
  Change in percent goal calories provided with enteral nutrition , measured percent of calorie provided with enteral nutrition from the estimated goal.
Change in percent goal proteins provided with enteral nutrition | Baseline, 12 weeks
  Change in percent goal proteins provided with enteral nutrition , measured percent of protein provided with enteral nutrition from the estimated goal.
Change in tube feeding tolerance | Baseline, 12 weeks
  Change in tolerance to tube feeding, measured by follow up questionnaire about symptoms of GI intolerance; namely, diarrhea, constipation, abdominal(stomach/tummy/belly) pain or discomfort, nausea and vomiting. The scale used will asses the frequency of these symptoms using the following terms: not at all, rarely, sometimes, often, and very often with not at all being least frequent and very often being most frequent presence of the concerning symptom.
Change in hand grip strength | Baseline, 12 weeks
  Change in hand grip strength, measured by dynamometer.
Change in diabetes medications | Baseline, 12 weeks
  Change in diabetes medications, measured by capturing any change in diabetes medications (when applicable) in terms of new medications added, or discontinuation or change in doses of current medications.
Change in anti-hypertensive medications | Baseline, 12 weeks
  Change in hypertension medications, measured by capturing any change in hypertension medications (when applicable) in terms of new medications added, or discontinuation or change in doses of current medications.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials